CLINICAL TRIAL: NCT02086981
Title: The DETEcT Study - Delirium in Elderly paTiEnts Admitted to Trauma
Acronym: DETEcT
Status: Completed | Type: Observational
Sponsor: Azienda Ospedaliero-Universitaria Careggi (Other)
Responsible Party: Principal Investigator, Alessandro Cartei, MD, Medicina Interna per la Gestione Pre e Postoperatoria Traumatologica e del Percorso Neuromotorio, Azienda Ospedaliero-Universitaria Careggi
Other Study IDs: OSS.13.070; OSS.13.070 (Other: Local Ethical Committee)
Record Dates: First submitted 2014-02-22; First posted 2014-03-14 (Estimated); Last update posted 2015-12-29 (Estimated); Status verified 2015-12

CONDITIONS: Delirium; Bone Fractures; Multiple Trauma
MeSH Terms: conditions — Delirium; Fractures, Bone; Multiple Trauma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No

SUMMARY:
Primary objectives are to define incidence and prevalence of Delirium in an elderly population admitted to the Department of Orthopedics and Traumatology and, in the postoperative phase, in the high Dependency Unit as well as to determine the presence of risk factors. Secondary objectives are to determine mean hospital stay, rates of complications as well as in-hospital mortality and at 1-3 and 12 months after discharge, functional recovery and cognitive outcomes at 1, 3 and 12 moths follow-up.

DETAILED DESCRIPTION:
The aging of population as well as the increased life expectancy put progressively urgent demands about the adequacy of the level of care provided in a hospital environment to ensure clinical pathways tailored on the needs of each individual patient. On the other hand, the gradual evolution of Health Care systems to care for the acute, with increasing levels of specialization often technologically driven, cannot and must not neglect these aspects of personalization of care protecting the elderly "frail" patient, because of its intrinsic characteristics. In such a context, evaluation of frailty undertakes not only the meaning of prevention and promotion of quality of life but it takes in account important issues for patient's safety and the economic weight it entails. Delirium (acute confusional state) is a complex syndrome which frequently occurs in the elderly hospitalized population. Development of Delirium is associated with negative outcomes such as a longer hospital stay, a higher rate of complications, cognitive and functional decline, loss of independence, institutionalization, and, ultimately, death. For skilled healthcare professionals, on the other hand, it represents a challenging condition because a prompt and accurate diagnosis with the introduction of all those prevention and non-pharmacological measures may reduce the incidence, severity and/or duration of Delirium and improve functional recovery. Therefore the meaning of conducting such an observational study is also to provide evidence of patients' needs and address the on-ground educational aspect for healthcare professionals in a daily practice. The purposes of the study are to determine the incidence and prevalence (before and after surgery) of Delirium in an elderly population admitted to the Department of Orthopedics and Traumatology and in the High Dependency Unit in the postoperative phase as well as to determine the risk factors for developing such a condition. Secondary objectives are mean hospital stay, rates of complications as well as in-hospital mortality and at 1, 3 and 12 months after discharge, functional recovery and cognitive outcomes at 1, 3 and 12 months follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Patients with any medical condition with an age of 65 years and older

Exclusion Criteria:

* Impossibility to give an informed consent; refusal

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Patients admitted to the Department of Orthopedics and Traumatology and in the High Dependency Unit in the postoperative phase
Sampling Method: Non-Probability Sample
Enrollment: 672 (Actual)
Dates: Start 2014-02; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Prevalence of Delirium, its association with risk factors and their prognostic value | At hospital admission
  Patients are evaluated on admission with:
  * IqCode
  * Katz Index of Independence in Activities of Daily Living (ADL)
  * The Lawton Instrumental Activities of Daily Living (IADL) Scale
  * The Barthel Index for Mobility
  * The Confusion Assessment Method (CAM)
  * The 4AT Scale
  * Presence of Risk Factors
Incidence of Delirium, its association with risk factors and their prognostic value | At hospital admission and for the next 48 hours
  Detection of any change in clinical condition. Patients are evaluated with:
  * The Confusion Assessment Method (CAM)
  * The 4AT Scale
Incidence of Delirium, its association with risk factors and their prognostic value | After surgery and for the next 48 hours
  Detection of any change in clinical condition. Patients are evaluated with:
  * The Confusion Assessment Method (CAM)
  * The 4AT Scale

SECONDARY OUTCOMES:
Mortality rates | In-Hospital
Mortality rates | At 1,3 and 12 months follow-up
Mean Hospital Stay | In-Hospital
Clinical Complications | In-Hospital
Changes in functional capabilities | At 1, 3 and 12 months follow-up
  Patients are evaluated with:
  * Katz Index of Independence in Activities of Daily Living (ADL)
  * The Lawton Instrumental Activities of Daily Living (IADL) Scale
  * The Barthel Index for Mobility

OTHER OUTCOMES:
Variations of serum cystatin C as a marker of glomerular filtration rate and its association with the development of Delirium | At hospital admission and on the fifth day of hospitalization

CONTACTS AND LOCATIONS:
Overall Officials: Marco Mannucci, MD, Study Director — Azienda Ospedaliero-Universitaria Careggi; Alessandro Cartei, MD, Principal Investigator — Azienda Ospedaliero-Universitaria Careggi
Locations (1):
- C.T.O. Azienda Ospedaliero-Universitaria Careggi, Florence, Italy